CLINICAL TRIAL: NCT05237609
Title: Effect of Muscle Strengthening on the Incidence of Psychomotor Disadaptation Syndrome After a Fall in Elderly Persons
Brief Title: Effect of Muscle Strengthening on the Incidence of Psychomotor Disadaptation Syndrome in Elderly Persons
Acronym: RM-SDP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 8455
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Psychomotor Disadaptation Syndrome; Post-fall Syndrome
Keywords: elderly person; muscle strengthening
MeSH Terms: interventions — Rehabilitation; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rehabilitation with muscle strengthening + Oral Nutritional Supplements (Experimental): Participants will receive weekly physical therapy sessions for 20 weeks, during their usual follow-up at the day hospital. In addition to the standard treatment, muscle strengthening exercises using elastic bands of varying resistance will be performed. These sessions can be completed by a muscle strengthening session at home during the week, given by a private physiotherapist according to the indication given by a doctor taking care of the patient, during and outside the periods of follow-up at the day hospital. In addition to muscle strengthening, participants will receive a systematic protein intake via Oral Nutritional Supplements (ONS) to improve muscle strength. Compliance with these oral nutritional supplements will be monitored by means of a booklet filled in by the patient or his entourage.
  Interventions: Dietary Supplement: rehabilitation with muscle strengthening + Oral Nutritional Supplements
- standard rehabilitation +/- Oral Nutritional Supplements (Active Comparator): The participants in the control group will receive the usual care at the day hospital, i.e. a rehabilitation program focused on the prevention of falls. The prescription of ONS will be made on a case-by-case basis by the day hospital's physician. If participants require follow-up by a physiotherapist at home, sessions will be prescribed.
  After the treatment, participants in the experimental group will be advised to continue the muscle strengthening sessions independently at least once a week. All participants, regardless of their group, who require follow-up by a physiotherapist will benefit from it.
  Interventions: Other: rehabilitation with muscle strengthening

INTERVENTIONS:
Dietary Supplement: rehabilitation with muscle strengthening + Oral Nutritional Supplements — Combination of protein intake and muscle strengthening exercises for the improvement of walking capacities, patients in the experimental group
  Arms: rehabilitation with muscle strengthening + Oral Nutritional Supplements
Other: rehabilitation with muscle strengthening — Physical activity with only muscle strengthening
  Arms: standard rehabilitation +/- Oral Nutritional Supplements

SUMMARY:
The post-fall syndrome or psychomotor disadaptation syndrome can be considered as a complication of a fall and can lead to a total loss of autonomy. This syndrome remains little studied, despite its important frequency in acute geriatric services or geriatric rehabilitation care, and despite its recognized seriousness. Decreased grip strength seems to be a risk factor for psychomotor disadaptation syndrome in after a fall, which is why we hypothesize that muscle strengthening adapted to the elderly subject would limit the appearance of this syndrome. By limiting this risk, it would reduce complications such as loss of functional independence, but also reduce the number and duration of hospitalization of elderly patients.

DETAILED DESCRIPTION:
The participants will be referred by the attending physicians, the physicians of the emergency department or the conventional hospitalization services of the University Hospital of Strasbourg to the "fall" consultation held at the Robertsau Hospital in geriatrics. Participants will be evaluated by experienced geriatricians. As part of their routine care, participants will receive

* A medical assessment
* Medical history,
* Significant medical history and assessment of comorbidities using the Charlson score,
* Medications and ONS (Oral Nutritional Supplements),
* Lifestyle,
* Complete clinical examination with orthostatic hypotension test and ECG,
* Cognitive assessment with MMSE,
* Retrieval of latest imaging and biology results.

If and only if the subject has signed his consent, the following measurements will be performed:

* Grip strength using a manometer,
* Gait assessment (gaitride® treadmill).

As in current practice, the patient will then be referred by the investigator to the ABRAPA day hospitals. They will then receive adapted management at the day hospital within 4 to 6 weeks of inclusion.

The intervention will be randomized:

- Experimental group: rehabilitation with muscle strengthening + ONS

Participants will receive weekly physical therapy sessions for 20 weeks, during their usual follow-up at the day hospital. In addition to the standard treatment, muscle strengthening exercises using elastic bands of varying resistance will be performed. These sessions can be completed by a muscle strengthening session at home during the week, given by a private physiotherapist according to the indication given by a doctor taking care of the patient, during and outside the periods of follow-up at the day hospital. In addition to muscle strengthening, participants will receive a systematic protein intake via Oral Nutritional Supplements (ONS) to improve muscle strength. Compliance with these oral nutritional supplements will be monitored by means of a booklet filled in by the patient or his entourage.

- Control group: standard rehabilitation +/- ONS

The participants in the control group will receive the usual care at the day hospital, i.e. a rehabilitation program focused on the prevention of falls. The prescription of ONS will be made on a case-by-case basis by the day hospital's physician. If participants require follow-up by a physiotherapist at home, sessions will be prescribed.

After the treatment, participants in the experimental group will be advised to continue the muscle strengthening sessions independently at least once a week. All participants, regardless of their group, who require follow-up by a physiotherapist will benefit from it.

Follow-up will take place for 2 years with data collected every 4 months from the inclusion visit via telephone calls to participants and their families, to the treating physician. A new medical evaluation is planned at 1 year, based on the same model as the screening visit, except for grip strength.

Participants will have a second cycle of 20 sessions at the day hospital in their respective group at the beginning of the second year of follow-up.

The end-of-study visit will take place 2 years after the inclusion visit in the same way as the 1-year visit.

The data collected will concern the onset of psychomotor maladjustment syndrome, the number of falls, severe falls, assessment of functional autonomy during follow-up, hospitalizations, hospitalizations for falls, entry into an institution, deaths from any cause, post-fall deaths.

ELIGIBILITY:
Inclusion criteria:

* Subject over 70 years of age at the time of signing the consent, with no upper limit,
* History of a fall,
* Subject affiliated with a social health insurance plan, beneficiary or beneficiary's assistant
* Subject able to understand the objectives and risks of the research and to give dated and signed informed consent.

Exclusion criteria:

* Osteoarticular limitations compromising muscle strengthening,
* Unstabilized cardiac pathologies,
* Unstabilized chronic pathologies,
* Unstabilized ventricular and supraventricular rhythm disorders or ECG abnormalities at the inclusion visit,
* Swallowing disorders (CNO)
* Acute coronary syndrome < 1 month,
* Unstabilized or oxygen-dependent respiratory failure,
* Cognitive impairment compromising muscle strengthening achievement (MMSE<22/30),
* Evolving cancers,
* Subject under guardianship or curatorship,
* Severe malnutrition,
* Severe functional limitation.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of psychomotor disadaptation syndrome | 2 years
  The primary endpoint will be the incidence of psychomotor disadaptation syndrome after a fall in subjects over 70 years of age who are receiving or not receiving adapted muscle strengthening. The determination of the psychomotor disadaptation syndrome is clinical and includes retropulsion, fear of falling, fear of verticality, oppositional hypertonia or an abrupt break with the previous functional state without obvious organic cause. It can be identified after of a fall by the family, by the nurses and physiotherapists in charge of the participants, by the doctors and physiotherapists of the HDJ, by their GP, by the emergency physicians if the patient is referred to the emergency room, by the hospital doctors in case of hospitalization, and will be identified during the visits at 1 and 2 years and during the telephone calls every 4 months.

SECONDARY OUTCOMES:
Incidence of psychomotor disadaptation syndrome complications following a fall | 2 years
  the number of falls, repeat falls (≥ 2 falls in a 12-month period)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gériatrie aigue - CHU de Strasbourg - France, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided